CLINICAL TRIAL: NCT04972669
Title: The Study of Electrical Acupuncture Stimulation Therapy for Postprostatectomy Incontinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Executive officer of Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IUNU-PC-105
Record Dates: First submitted 2021-07-09; First posted 2021-07-22 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-11

CONDITIONS: Postprostatectomy Incontinence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Sham Comparator): sham electroaupuncture
  Interventions: Device: sham Acupuncture
- experimental group (Experimental): Electroaupuncture
  Interventions: Device: Electrical Acupuncture Stimulation

INTERVENTIONS:
Device: Electrical Acupuncture Stimulation — Participants received acupuncture at bilateral Baliao. After skin disinfection, sterile adhesive pads were placed on bilateral Baliao, and acupuncture needles were inserted through the adhesive pads. Following needle insertion, small, equal manipulations of twirling, lifting, and thrusting were performed on all needles to reach de qi. Electrodes from the electroacupuncture apparatus were attached transversely to the needle handles. The electroacupuncture stimulation lasted for 30 minutes with a continuous wave of 2-15 Hz. Participants received 3 treatment sessions per week (ideally every other day) for 6 consecutive weeks, 18 sessions in total.
  Arms: experimental group
Device: sham Acupuncture — Participants received sham acupuncture at locations one inch besides bilateral Baliao without needle insertion. Electrodes from the electroacupuncture apparatus were attached transversely to the needle handles. The electroacupuncture stimulation lasted for 30 minutes with a continuous wave of 2-15 Hz. Participants received 3 treatment sessions per week (ideally every other day) for 6 consecutive weeks, 18 sessions in total.
  Arms: control group

SUMMARY:
More than 50% patients underwent prostatectomy suffered from postoperative incontinence, and the effect of pelvic floor muscle training is very limited. Electrical acupuncture stimulation therapy has been demonstrated to work on other kinds of Urinary Incontinence. Before this trial, the researchers have conducted pre-experiments where electrical acupuncture stimulation therapy was conducted for few postprostatectomy Incontinence patients. On the basis of the preliminary work, this prospective, random control research aims to verify the safety and effectiveness of electroacupuncture in the treatment of postprostatectomy Incontinence.

ELIGIBILITY:
Inclusion Criteria:

* localized prostate cancer (stage: cT1-cT2, N0, M0)
* 4-6weeks after prostatectomy
* postprostatectomy prostate specific antigen (PSA) test below cured level
* incontinence one month after surgery
* ECOG score:0-1

Exclusion Criteria:

* history of neoadjuvant hormonal therapy
* history of transurethral resection of the prostate (TUPR)
* history of operation on pelvis
* history of incontinence before prostatectomy

Max Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 110 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Continence rate after 6 weeks of treatment | 3 years

SECONDARY OUTCOMES:
change of urine pad quantity for 24 hours after 4 courses compared with baseline | 3 years
change of weight in kilograms of urine pad for 24 hours after 6 courses compared with baseline | 3 years
changes of The expanded prostate cancer index composite(EPIC) score after 4-6 courses compared with baseline | 3 years
Long-term urinary continence recovery | 3 year
  time from randomization to urinary continence

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Niu J, Wang Y, Wang Y, Shi J, Liang J, Zhao X, Xu T, Guo H, Qiu X. Electroacupuncture in Patients With Early Urinary Incontinence After Radical Prostatectomy: A Randomized Clinical Trial. JAMA Netw Open. 2025 Sep 2;8(9):e2534491. doi: 10.1001/jamanetworkopen.2025.34491. PMID 41026492